CLINICAL TRIAL: NCT03965598
Title: Study on Predictiors and Mechanism of Conversion to Psychosis in Individuals at Ultra-high Risk Group
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Xiangya Hospital of Central South University (Other)
Collaborators: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xiaogang Chen, Professor, Second Xiangya Hospital of Central South University
Other Study IDs: 81871056
Record Dates: First submitted 2019-05-26; First posted 2019-05-29 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Ultra-high risk for psychosis; Predictors; Pathogenesis
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Genomic DNA and RNA will be extracted respectively from white blood cells in peripheral blood.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ultra-high risk for psychosis (UHP): Ultra-high risk for psychosis (UHP) is defined as individuals at the prodromal stage of schizophrenia.
  Inclusion Criteria: age of 13-30 years; meet the diagnostic criteria of COPS prodromal syndrome by SIPS clinical interviews; have not received any psychiatric medication; be in good health, without major mental illness or physical illness; normal intelligence, can be operated on a clinical scale; volunteer to participate in the study and sign the written consent form.
  Exclusion criteria: exclusion of current or previous psychiatric disorders by SCID interview; meet the diagnostic criteria for substance abuse and substance dependence in DSM-IV; contraindications for MRI; pregnant or lactating women.
- Healthy controls: Inclusion Criteria: the gender, age, and education level of the group are matched with the Ultra-high risk group; 13 to 30 years old; right-handed; no history of mental illness; no mental disorder consistent with DSM-IV diagnostic criteria within two or three generations; No contraindications for MRI; volunteer to participate in the study and sign the written consent form.
  Exclusion criteria: history of disturbance of consciousness over 5 minutes; history of brain organic disease or head injury; history of alcohol and drug dependence; history of coma; history of endocrine disease; abnormity in examination of blood, heart, liver, or renal function; pregnant or lactating women.

SUMMARY:
Considering the complex pathological mechanism and the poor treatment outcomes of schizophrenia, early detection and intervention gradually become the key work for the foundational and clinical research in schizophrenia. Ultra-high risk for psychosis (UHP) is defined as individuals at the prodromal stage of schizophrenia. Early intervention in individual at UHP can effectively delay or even prevent the development of the illness. Long-term longitudinal studies suggested that there are clinical outcomes in people at UHP. Nearly 1/3 of individuals at UHP may be naturally relieved without any intervention, about 1/3 of individuals at UHP will remain at the prodromal stage of schizophrenia, and only 1/3 individuals at UHP will eventually develop schizophrenia. In this regard, it will cause adverse effects on false positive individuals if they accept clinical intervention. Unfortunately, it is difficult to accurately predict which individuals at UHP will make a transition to frank illness. To solve this issue, we explore the association between baseline brain structural and functional networks, methylation modifications, gene expression, neurocognitive function and the clinical outcomes of UHP individuals, and to identify the potential biological and clinical predictors for the long-term outcomes in the individuals at UHP. In addition, we also detect the changes of brain structure and function, methylation status and gene expression in individuals at UHP during follow-up, and further to investigate the etiology and pathogenesis of schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* 1. age of 13-30 years;
* 2. meet the diagnostic criteria of COPS prodromal syndrome by SIPS clinical interviews;
* 3. have not received any psychiatric medication;
* 4. be in good health, without major mental illness or physical illness;
* 5. normal intelligence, can be operated on a clinical scale;
* 6. volunteer to participate in the study and sign the written consent form.

Exclusion Criteria:

* 1. exclusion of current or previous psychiatric disorders by SCID interview;
* 2. meet the diagnostic criteria for substance abuse and substance dependence in DSM-IV;
* 3. contraindications for MRI;
* 4. pregnant or lactating women.

Ages: 13 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Ultra-high risk for psychosis (UHP) is defined as individuals at the prodromal stage of schizophrenia.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-11-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Conversion to psychosis. | Two years.
  Conversion is operationalized as the criteria of POPS (Presence of Psychotic Symptoms in SIPS/SOPS). Subjects have to demonstrate at least one psychotic level symptom (rated a '6') on at least one of the five P(Positive) symptoms (P1, unusual thought content; P2, suspiciousness; P3, grandiosity; P4, perceptual abnormalities; and P5, disorganized communication), with either sufficient frequency and duration or at a level that is disorganizing or dangerous.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaogang Chen, Ph.D, Principal Investigator — Professor
Locations (1):
- The 2nd Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] He Y, Kosciolek T, Tang J, Zhou Y, Li Z, Ma X, Zhu Q, Yuan N, Yuan L, Li C, Jin K, Knight R, Tsuang MT, Chen X. Gut microbiome and magnetic resonance spectroscopy study of subjects at ultra-high risk for psychosis may support the membrane hypothesis. Eur Psychiatry. 2018 Sep;53:37-45. doi: 10.1016/j.eurpsy.2018.05.011. Epub 2018 Jun 2. PMID 29870894
- [Background] He Y, Li Z, Ma X, Yuan L, Ouyang L, Tang J, Tsuang MT, Chen X. Olfactory and cognitive functions in Chinese individuals at clinical high risk for psychosis. Psychiatry Res. 2019 Feb;272:51-53. doi: 10.1016/j.psychres.2018.12.074. Epub 2018 Dec 14. PMID 30579181
- [Background] He Y, Yuan L, Li Z, Zhou Y, Ma X, Ouyang L, Chen X. Plasma protein levels of brain-derived neurotrophic factor pathways and their association with cognitive performance in patients with clinical high risk for psychosis and first episode psychosis. Schizophr Res. 2019 Apr;206:460-461. doi: 10.1016/j.schres.2018.11.016. Epub 2018 Nov 28. No abstract available. PMID 30503369
- [Derived] Wang Y, Ouyang L, Fan L, Zheng W, Li Z, Tang J, Yuan L, Li C, Jin K, Liu W, Chen X, He Y, Ma X. Functional and structural abnormalities of thalamus in individuals at early stage of schizophrenia. Schizophr Res. 2024 Sep;271:292-299. doi: 10.1016/j.schres.2024.07.045. Epub 2024 Jul 29. PMID 39079406
- [Derived] Ma X, Yang WFZ, Zheng W, Li Z, Tang J, Yuan L, Ouyang L, Wang Y, Li C, Jin K, Wang L, Bearden CE, He Y, Chen X. Neuronal dysfunction in individuals at early stage of schizophrenia, A resting-state fMRI study. Psychiatry Res. 2023 Apr;322:115123. doi: 10.1016/j.psychres.2023.115123. Epub 2023 Feb 20. PMID 36827856